CLINICAL TRIAL: NCT03082079
Title: Long Outcome of Endoscopic Submucosal Dissection for Small Gastrointestinal Stromal Tumors (<2cm) :a Randomized Controlled Trial
Brief Title: Long Outcome of Endoscopic Submucosal Dissection for Small Gastrointestinal Stromal Tumors (<2cm)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LC2016YM002
Record Dates: First submitted 2017-03-01; First posted 2017-03-17 (Actual); Last update posted 2017-05-16 (Actual); Status verified 2017-02

CONDITIONS: GIST
Keywords: GIST; ESD

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESD group (Experimental): Patient in this group undergo ESD for GIST, and regular follow-up are carried out for these patients on 72 ±3h,7±2d,14±2d,3 month,6 month,1 year,2 year,3 year,4 year,5 year after the treatment. The investigators record the success rate of operation,en bloc resection,operation time,complication rate,hospitalization days,hospitalization expenses,pathology results and tumor recurrence rate.
  Interventions: Procedure: ESD
- Follow-up group (No Intervention): Patient in this group are given no intervention,the investigators record the tumor size and EUS features of the first endoscopic examination.Regular follow-up are carried out for these patients on 3 month,6 month,1 year,2 year,3 year,4 year,5 year after this check.Then,tumor size and EUS features of each time are collected accurately.

INTERVENTIONS:
Procedure: ESD — Patient in ESD group undergo ESD for GIST, and regular follow-up are carried out for these patients on 72 ±3h,7±2d,14±2d,3 month,6 month,1 year,2 year,3 year,4 year,5 year after the treatment. The investigators record the success rate of operation,en bloc resection,operation time,complication rate,hospitalization days,hospitalization expenses,pathology results and tumor recurrence rate
  Arms: ESD group

SUMMARY:
Data are currently insufficient to guide the management of very small gastrointestinal stromal tumors（GISTs）（< 2 cm) discovered incidentally on endoscopy,this study is designed to collect the medical records of patients in different treatment group with long-term follow-up data,and attempts to evaluate the usefulness of regular endoscopic ultrasound（EUS）surveillance and the necessity,safety and feasibility of endoscopic submucosal dissection（ESD）for small GISTs,thus provide evidence for the revision of the guideline.

DETAILED DESCRIPTION:
OBJECTION:to evaluate the usefulness of regular endoscopic ultrasound（EUS） surveillance and the necessity,safety and feasibility of endoscopic submucosal dissection（ESD） for small GISTs(<2cm),thus providing evidences for the revision of the guideline.

OUTLINE:This is a randomized controlled trial. Eligible patients are divided into 2 group with 45 in each.The experimental group undergo ESD for GISTs,while the investigators do no treatment to the control group.Then,the 2 groups will be follow up for 5 years.All data are analysed with the Statistical Product and Service Solutions（SPSS）statistical software.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female chinese patients of 18-70 years old.
2. Patients with very small gastric GISTs (< 2 cm) with no high-risk EUS features.
3. Patients voluntarily join this study with informed consents.

Exclusion Criteria:

1. Patients with the tumors involving the serosa layer or grow outside the lumen obviously that are not eligible for endoscopic treatment.
2. Patients with distant metastasis on computed tomography(CT)scan.
3. patients with an extremely poor general condition or a very short life expectancy.
4. Patients presenting with severe gastrointestinal tract bleeding that require immediate surgery.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2017-06-01 (Estimated); Primary Completion 2021-08-01 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | 5 years
  It is the time that passes from a patient is enrolled in this clinical trial to the date on which disease "progresses" or the date on which the patient dies, from any cause.

SECONDARY OUTCOMES:
tumor recurrence rate | 5 years
  The proportion of the total number of patients with recurrence of each grop, which confirmed by endoscopic and other imaging data during follow-up.
success rate of operations | At surgery
  The proportion of the total number of patients with GISTs been successfully resected of each group.
Tumor progression rates | 5 years
  The proportion of the total number of patients with tumor continuing to increase of each group.
Operation time | At surgery
  It is the time that passes from ESD beginning to complete resection of the tumors.
Peri-operative bleeding | At surgery
  The amount of bleeding during operation.
Complications rate | At surgery
  Complications including bleeding and perforation.
Duration of hospitalization and the total hospital costs | through the whole recovery, an average of 10 days
  length of hospital stay and all costs related to the operations and examinations and the period of hospitalization.
Histological curative resection | At surgery
  Histological curative resection is defined as complete tumor removal which confirmed by pathological assessment of resected tissue
patient satisfaction scores | 5 years
  We administer questionnaires to each patients,and invite them to score for this treatment or examination.

CONTACTS AND LOCATIONS:
Overall Officials: yue li, Doctor, Study Chair — Nanfang Hospital, Southern Medical University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Davila RE, Faigel DO. GI stromal tumors. Gastrointest Endosc. 2003 Jul;58(1):80-8. doi: 10.1067/mge.2003.317. No abstract available. PMID 12838226
- [Background] Siow SL, Mahendran HA, Wong CM. Laparoscopic transgastric resection for intraluminal gastric gastrointestinal stromal tumors located at the posterior wall and near the gastroesophageal junction. Asian J Surg. 2017 Sep;40(5):407-414. doi: 10.1016/j.asjsur.2015.12.001. Epub 2016 Feb 24. PMID 26922628
- [Background] Reichardt P. [Soft tissue sarcomas and gastrointestinal stromal tumors]. Internist (Berl). 2016 Mar;57(3):245-56. doi: 10.1007/s00108-016-0021-2. German. PMID 26907871
- [Background] Ucar AD, Oymaci E, Carti EB, Yakan S, Vardar E, Erkan N, Mehmet Y. Characteristics of Emergency Gastrointestinal Stromal Tumor (GIST). Hepatogastroenterology. 2015 May;62(139):635-40. PMID 26897944
- [Background] Sornmayura P. Gastrointestinal stromal tumors (GISTs): a pathology view point. J Med Assoc Thai. 2009 Jan;92(1):124-35. PMID 19260254
- [Background] ESMO/European Sarcoma Network Working Group. Gastrointestinal stromal tumours: ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2014 Sep;25 Suppl 3:iii21-6. doi: 10.1093/annonc/mdu255. No abstract available. PMID 25210085
- [Background] Maghrebi H, Chebbi F, Makni A, Haddad A, Daghfous A, Fteriche F, Rebai W, Ksantini R, Jouini M, Kacem M, Ben Safta Z. Laparoscopic resection of gastric stromal tumors. Tunis Med. 2015 Oct;93(10):594-7. PMID 26895119
- [Background] Novitsky YW, Kercher KW, Sing RF, Heniford BT. Long-term outcomes of laparoscopic resection of gastric gastrointestinal stromal tumors. Ann Surg. 2006 Jun;243(6):738-45; discussion 745-7. doi: 10.1097/01.sla.0000219739.11758.27. PMID 16772777
- [Background] Nakamori M, Iwahashi M, Nakamura M, Tabuse K, Mori K, Taniguchi K, Aoki Y, Yamaue H. Laparoscopic resection for gastrointestinal stromal tumors of the stomach. Am J Surg. 2008 Sep;196(3):425-9. doi: 10.1016/j.amjsurg.2007.10.012. Epub 2008 May 7. PMID 18466871
- [Background] Matsuhashi N, Osada S, Yamaguchi K, Okumura N, Tanaka Y, Imai H, Sasaki Y, Nonaka K, Takahashi T, Futamura M, Yoshida K. Long-term outcomes of treatment of gastric gastrointestinal stromal tumor by laparoscopic surgery: review of the literature and our experience. Hepatogastroenterology. 2013 Nov-Dec;60(128):2011-5. PMID 24719942
- [Background] Demetri GD, von Mehren M, Antonescu CR, DeMatteo RP, Ganjoo KN, Maki RG, Pisters PW, Raut CP, Riedel RF, Schuetze S, Sundar HM, Trent JC, Wayne JD. NCCN Task Force report: update on the management of patients with gastrointestinal stromal tumors. J Natl Compr Canc Netw. 2010 Apr;8 Suppl 2(0 2):S1-41; quiz S42-4. doi: 10.6004/jnccn.2010.0116. PMID 20457867
- [Background] Deprez PH. Endoscopic diagnosis and treatment of upper gastrointestinal tumors. Endoscopy. 2011 Nov;43(11):966-70. doi: 10.1055/s-0031-1291427. Epub 2011 Nov 4. PMID 22057760
- [Background] Goto O, Uraoka T, Horii J, Yahagi N. Expanding indications for ESD: submucosal disease (SMT/carcinoid tumors). Gastrointest Endosc Clin N Am. 2014 Apr;24(2):169-81. doi: 10.1016/j.giec.2013.11.006. Epub 2014 Jan 25. PMID 24679229
- [Background] Meng Y, Cao C, Song S, Li Y, Liu S. Endoscopic band ligation versus endoscopic submucosal dissection and laparoscopic resection for small gastric stromal tumors. Surg Endosc. 2016 Jul;30(7):2873-8. doi: 10.1007/s00464-015-4571-5. Epub 2015 Oct 21. PMID 26490768
- [Background] Bang CS, Baik GH, Shin IS, Suk KT, Yoon JH, Kim DJ. Endoscopic submucosal dissection of gastric subepithelial tumors: a systematic review and meta-analysis. Korean J Intern Med. 2016 Sep;31(5):860-71. doi: 10.3904/kjim.2015.093. Epub 2016 Feb 22. PMID 26898597
- [Background] Cho JW; Korean ESD Study Group. Current Guidelines in the Management of Upper Gastrointestinal Subepithelial Tumors. Clin Endosc. 2016 May;49(3):235-40. doi: 10.5946/ce.2015.096. Epub 2016 Feb 22. PMID 26898512
- [Background] Zhang Q, Li Y, Meng Y, Bai Y, Cai JQ, Han ZL, Wang Z, Zhi FC, Liu SD. Should the Integrity of Mucosa Be Considered in Endoscopic Resection of Gastric Submucosal Tumors? Gastroenterology. 2016 Apr;150(4):822-4.e9. doi: 10.1053/j.gastro.2016.01.040. Epub 2016 Feb 11. No abstract available. PMID 26874075